CLINICAL TRIAL: NCT05497609
Title: The Muscle in Children Cerebral Palsy - Longitudinal Exploration of Microscopic Muscle Structure in Gastrocnemius and Biceps Brachii During Two Years of Care as Usual, Including Training With Botulinum Toxin Injections as Adjuvant Therapy.
Brief Title: The Muscle in Children With Cerebral Palsy - Longitudinal Exploration of Microscopic Muscle Structure.
Acronym: CPBiopsyBTX
Status: Recruiting | Type: Observational
Sponsor: Eva Ponten (Other Government)
Responsible Party: Sponsor-Investigator, Eva Ponten, MD PhD Ass Prof, Region Stockholm
Organization: Region Stockholm (Other Government)
Other Study IDs: BTX muskel CP
Record Dates: First submitted 2022-07-27; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy; Muscle Contraction; Muscle Spasticity
Keywords: Cerebral Palsy; Upper Limb; Lower Limb; Muscle Biopsy; Botulinum Toxin Type A
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Percutaneous muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention. Care as ususal — No intervention

SUMMARY:
Cerebral palsy (CP) is a motor impairment due to a brain malformation or a brain lesion before the age of two. Spasticity, hypertonus in flexor muscles, dyscoordination and an impaired sensorimotor control are cardinal symptoms. The brain lesion is non-progressive, but the flexor muscles of the limbs will during adolescence become relatively shorter and shorter (contracted), forcing the joints into a progressively flexed position. This will worsen the positions of already paretic and malfunctioning arms and legs. Due to bending forces across the joints, bony malformations will occur, worsening the function even further. Since about 25 years a combination treatment with intramuscular botulinum toxin injections, braces and training has had a tremendous and increasing popularity, although lasting long-term clinical advantage is not yet proven.

Muscle morphology of the biceps brachii and the gastrocnemius muscles:

* The hypothesis is that care as usual, i.e. training and splinting sessions with botulinum toxin as adjuvant treatment, will reduce (normalize) the expression of the fast fatigable myosin heavy chain MyHC IIx and increase the expression of developmental myosin, as a possible sign of growth. As the biceps in the arm is used irregularly and voluntarily, and the gastrocnemius is activated during automated gait, the adaptations of those muscles will be different. Methods: Baseline muscle biopsies: Percutaneous biopsies are taken just before the first intramuscular botulinum toxin injection is given. The doses and the intervals for the botulinum toxin treatment will follow clinical routines. Biopsies 4-6 months, 12 months and 24 months after the first botulinum toxin injection: The exact same procedure as above will be performed, but the biopsies will be taken 2 cm distant, medial or lateral, from previous biopsy sites
* Significance:. More knowledge is warranted regarding the actual molecular process in the muscle leading to a contracture, and its relation to the constant communication with the injured central nervous system. This study will give answers that could result in new, early prophylactic treatment of joint movement restrictions and motor impairment in children with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a motor impairment due to a brain malformation or a brain lesion before the age of two. Spasticity, hypertonus in flexor muscles, dyscoordination and an impaired sensorimotor control are cardinal symptoms. The brain lesion is non-progressive, but the flexor muscles of the limbs will during adolescence become relatively shorter and shorter (contracted), forcing the joints into a progressively flexed position. This will worsen the positions of already paretic and malfunctioning arms and legs. Due to bending forces across the joints, bony malformations will occur, worsening the function even further. Currently, the initial treatment of choice is the use of braces, which diminishes the shortening somewhat. Since about 25 years a combination treatment with intramuscular botulinum toxin injections, braces and training has had a tremendous and increasing popularity, although lasting long-term clinical advantage is not yet proven.

Muscle morphology of the biceps brachii and the gastrocnemius muscles:

• The hypothesis is that care as usual, i.e. training and splinting sessions with botulinum toxin as adjuvant treatment, will reduce (normalize) the expression of the fast fatigable myosin heavy chain MyHC IIx and increase the expression of developmental myosin, as a possible sign of growth. As the biceps in the arm is used irregularly and voluntarily, and the gastrocnemius is activated during automated gait, the adaptations of those muscles will be different. Methods: Baseline muscle biopsies: Percutaneous biopsies from the biceps brachii and the gastrocnemius muscles are taken just before the first intramuscular botulinum toxin injection is given. The doses and the intervals for the botulinum toxin treatment will follow clinical routines. Training of the leg and arm will after the injections be performed with the help of physiotherapists and occupational therapists. Biopsies 4-6 months, 12 months and 24 months after the first botulinum toxin injection: The exact same procedure as above will be performed, but the biopsies will be taken 2 cm distant, medial or lateral, from previous biopsy sites. The muscle specimens are snap frozen and stored at -80°C until analyzed. The expression of different myosin heavy chain (MyHC) isoforms is assessed by using the monoclonal antibodies (mAb) N2.261, mAb A4.840 against slow MyHC I, mAb F1.652 against embryonic MyHC, and mAb NCL-MHCn against fetal (=neonatal) MyHC)(Tiger, Champliaud et al. 1997; Wewer, Thornell et al. 1997). Satellite cells will be identified with mAb against N-CAM (neural cell adhesion molecule). The fibers are typed according to the content of MyHCs.

Significance: Children with cerebral palsy have a motor impairment and progressive contractures that we often treat late; when tendon and bony surgery are the only options to realign the joints. Our aim is to treat the muscles early, so that the contractures and the bony malformations won't occur in the first place. Training and splints, with botulinum toxin as adjuvant treatment, is a very popular regime with this aim, but the long-term effect on muscle tissue and function is not yet known. This study will elucidate the effect during a 2-year period, and no such studies have yet been published. More knowledge is warranted regarding the actual molecular process in the muscle leading to a contracture, and its relation to the constant communication with the injured central nervous system. This study will give answers that could result in new, early prophylactic treatment of joint movement restrictions and motor impairment in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy, Aquired Brain Injury

Exclusion Criteria:

* Progressive neural disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cerebral palsy and aquired brain injury who, as a part of care as usual, gets botulinum toxin injections in muscles. Children are recruited consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-01-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Muscle fiber area | Biopsies are collected and stored in -80° freezer and then analyzed. Analyses will take place up to 20271215
  um2, square micrometers, measured on specimens
Muscle fiber types based on myosin heavy chain isoforms | Biopsies are collected and stored in -80° freezer and then analyzed. Analyses will take place up to 20271215
  Percentage of all fibers
Extracellular matrix, area | Biopsies are collected and stored in -80° freezer and then analyzed. Analyses will take place up to 20271215
  um2, square micrometers, measured on specimens
Capillaries per fiber area | Biopsies are collected and stored in -80° freezer and then analyzed. Analyses will take place up to 20271215
  number of capillaries/um2
Mitochondria: NADH staining, morphology | Biopsies are collected and stored in -80° freezer and then analyzed. Analyses will take place up to 20271215
  Scoring 1, 2, 3

SECONDARY OUTCOMES:
Clinical assessment, contracture | At 0 months, 6 months, 12 months and 24 months
  °, degrees

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Pontén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided